CLINICAL TRIAL: NCT04322916
Title: Clinical Study With the RM Pressfit Vitamys Cup in Combination With a Mathys Stem
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mathys Ltd Bettlach (Industry)
Responsible Party: Sponsor
Other Study IDs: 20081020_Protocol_E_vitamys_V1
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Arthropathy of Hip; Hip Replacement
Keywords: Primary osteoarthritis; Secondary osteoarthritis; Inflammatory arthritis; Congenital dysplasia; Femoral head fracture
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RM Pressfit vitamys: Participants treated with a RM Pressfit vitamys hip cup in combination with a Mathys hip stem
  Interventions: Device: RM Pressfit vitamys

INTERVENTIONS:
Device: RM Pressfit vitamys — Implantation of a RM Pressfit vitamys hip cup

SUMMARY:
The purpose of the study is the evaluation of the clinical and radiological short- to long-term safety and performance of the RM Pressfit vitamys cup. The data will be used for an ongoing evaluation of the product safety and performance.

DETAILED DESCRIPTION:
Prospective multicenter follow-up study which examines the short- to long-term post-market clinical data on the safety and performance of the RM Pressfit vitamys cup. In total 675 participants in 9 clinics are included in this international multicenter study.

The primary endpoint of the study is the Harris Hip Score (HHS) 2 years after surgery.

The following parameters will be collected during the regular clinical and radiological follow-up: Harris Hip Score, radiographic evaluation and detection of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form (signed by participant and investigator)
* Primary implantation
* Age at inclusion: Between 18 and 95 years old
* Willing to participate in the follow-up

Exclusion Criteria:

* Missing Informed consent form
* Known or suspected non-compliance (e.g. drug or alcohol abuse)
* Enrollment of the investigator, his/her family, employees and other dependent persons
* Patient younger than 18 years old
* Revision surgery
* Presence of sepsis or malignant tumors
* Pregnancy

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: according to Eligibility Criteria
Sampling Method: Non-Probability Sample
Enrollment: 675 (Actual)
Dates: Start 2009-09-15 (Actual); Primary Completion 2012-03-28 (Actual); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score (modified after Haddad et al, 1990) | 2 years
  The primary endpoint of the study is the Harris Hip Score (HHS) 2 years after surgery. The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.

SECONDARY OUTCOMES:
Radiographic evaluation | 6-12 weeks - 10 years
  The second endpoint of interest is the occurence of osteolysis around the cup
Adverse Events | 6-12 weeks - 10 years
  Reporting of Adverse Events

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Afghanyar Y, Joser S, Tecle J, Drees P, Dargel J, Rehbein P, Kutzner KP. The concept of a cementless isoelastic monoblock cup made of highly cross-linked polyethylene infused with vitamin E: radiological analyses of migration and wear using EBRA and clinical outcomes at mid-term follow-up. BMC Musculoskelet Disord. 2021 Jan 23;22(1):107. doi: 10.1186/s12891-021-03981-8. PMID 33485345